CLINICAL TRIAL: NCT04679688
Title: Acıbadem University Medical Faculty Atakent Hospital IVF Unit
Brief Title: Comparison of Follicle Diameter on hCG Day and Follicle Diameters on OPU (Oocyte Pick up) Day and the Effect of Follicle Diameters on Embryo Development and Pregnancy Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: ATAKIVF
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: HCG Day Follicle Diameter, Reproduction Results
MeSH Terms: interventions — Pregnancy Outcome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: descriptive — Those who apply for IVF treatment and have an antral follicle number of 4-10 will be included in the treatment. The reason for including patients with this number of antral follicles in the study is to determine the follicle locations and to determine each growing follicle separately on the day of hCG and egg collection.
  Other Names: The effect of follicle diameters on embryo development and pregnancy outcomes.

SUMMARY:
Evaluation of follicle diameters on human chorionic gonadotrophin(hCG) day and oocyte pick up (OPU) day of follicles developing after gonadotropin treatment, the relationship between follicle diameter and maturation in oocytes obtained after OPU and its effect on pregnancy outcomes will be investigated. In order to make it easier to measure and enumerate the follicle diameters with the help of vaginal ultrasound, patients under 35 years of age with at most five follicles in any ovary and at least four follicles in both ovaries will be included in the study.

DETAILED DESCRIPTION:
In our study, patients with 5 and 10 follicles exceeding 11 mm will be included in order to define the follicles whose hCG day is measured more clearly on the day of OPU in patients with whom we performed controlled ovarian hyperstimulation for in vitro fertilisation(IVF). The localizations and diameters of these follicles in both ovaries will be drawn and the hCG day will be numbered and their measurements will be indicated. On the day of opu, the marked and numbered follicles will be measured, noted and aspirated one by one, the collected eggs will be followed in individually numbered culture dish and it will be evaluated whether they are mature or not prepared for microinjection. And mature oocytes will be followed in numbered culture dishes after microinjection. The relationship between hCG and OPU day follicle diameter will be evaluated by following the follicle diameter and follicle diameters on the day of egg collection, the relationship between the mature egg, the rate of reaching the blastocyst stage, the clinical pregnancy and live birth rates

Especially the relationship between mature egg and follicle diameter and the resulting clinical results may guide clinicians in practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patient group with at least 5 and at most 10 follicles in each ovary whose hCG day exceeds 11 mm,
2. Patient group with BMI below 30.

Exclusion Criteria:

1. PCO patient group,
2. Male factor group with severe OAT,
3. Patient group with endometriosis,
4. Patient group with PGD indication,
5. The group under the age of 40 and legally deserving of double embryo transfer

Ages: 23 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 15 months
  live birth rate of participants
Clinical pregnancy rate | 6 months
  clinical pregnancy rate of participants

SECONDARY OUTCOMES:
Oocyte maturation | 6 months
  Oocyte maturation rate of participants

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Acıbadem University Atakent Hospital, Istanbul, Küçükçekmece
  - Acibadem MAA University Atakent Hospital, Istanbul